CLINICAL TRIAL: NCT03648684
Title: Examining Expectancy Challenges to Prevent Nonmedical Prescription Stimulant Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Alison Looby, Assistant Professor, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20180620AL02017
Record Dates: First submitted 2018-07-05; First posted 2018-08-27 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Prescription Drug Abuse (Not Dependent)
Keywords: Nonmedical prescription stimulant use; Expectancy challenge; College students
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeine-Based Expectancy Challenge (Experimental): Participants will ingest caffeine under the guise of Adderall prior to completing tasks. They will engage in an expectancy challenge intervention designed to both challenge expectancies for prescription stimulants and promote safe caffeine use for cognitive/mood enhancement.
  Interventions: Behavioral: Caffeine-Based Expectancy Challenge
- Placebo-Based Expectancy Challenge (Placebo Comparator): Participants will ingest placebo under the guise of Adderall prior to completing tasks. They will engage in an expectancy challenge intervention designed to challenge expectancies for prescription stimulants.
  Interventions: Behavioral: Placebo-Based Expectancy Challenge
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Caffeine-Based Expectancy Challenge — Intervention to alter expectancies and encourage safe drug substitution (harm reduction plus expectancy modification)
  Arms: Caffeine-Based Expectancy Challenge
Behavioral: Placebo-Based Expectancy Challenge — Intervention to alter expectancies (expectancy modification only)
  Arms: Placebo-Based Expectancy Challenge

SUMMARY:
Nonmedical prescription stimulant use (NPS) is commonly reported among college students for cognitive enhancement purposes, though it is associated with numerous negative psychological and physical consequences. Despite increasingly high prevalence rates and widespread acknowledgement of the need for efficacious interventions, little is known regarding how to prevent or treat this behavior. An intervention that targets cognitive enhancement motives and expectancy effects related to NPS may be particularly effective in light of recent research purporting limited evidence for meaningful NPS-related cognitive improvements among individuals without legitimate attention deficits. The primary objective of this proposal is to examine the efficacy of an intervention that successfully prevents NPS among college students by modifying expectations for NPS-related effects, while at the same time providing alternative means of enhancing cognition and arousal. Participants will be 126 stimulant-naïve college students who report a combination of risk factors for NPS. They will be randomized to one of three treatment conditions: a placebo-based expectancy challenge intervention that solely aims to modify expectancies related to NPS, a caffeine-based expectancy challenge intervention that includes expectancy modification combined with a safer alternative for cognitive enhancement, or a control group. Multilevel mixed modeling and survival analyses will be used to 1) examine changes in NPS-related expectancy effects across a 6-month follow-up period, and 2) assess incidence of NPS over the follow-up period, respectively, across the three groups. It is hypothesized that both expectancy challenge interventions will successfully modify expectancies compared to the control group and that they will be maintained over the follow-up period. It is also expected that the caffeine-based intervention will most successfully prevent NPS through a combination of expectancy modification and encouraging safe use of caffeine rather than prescription stimulants to achieve desired outcomes. Mediational analyses will also be employed to assess whether changes in expectancy effects via the interventions are responsible for differences in initiation rates between groups. The results of this project will facilitate the development of larger-scale prevention efforts to target the high rate of NPS on college campuses.

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers
* Current undergraduate enrollment
* Prescription stimulant naive
* At-risk for nonmedical prescription stimulant use, defined by endorsement of 2+ risk factors: male sex OR white race, Greek involvement, GPA < 3.5, past two-week binge drinking, past-month marijuana
* Willingness to ingest Adderall in the laboratory
* Past-month caffeine use

Exclusion Criteria:

* Lifetime history of use of any prescription stimulant
* Current psychiatric diagnosis
* Current psychiatric medication use
* Smoking > 5 cigarettes daily or daily use of any other nicotine product
* History of cardiac problems, diabetes, or regular hypoglycemia
* Current pregnancy or breastfeeding
* History of adverse reactions to caffeine

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Prescription Stimulant Expectancy Modification | 7 months
  This will be assessed via changes on the Prescription Stimulant Expectancy Questionnaire-II. This scale includes 4 subscales, each of which will be assessed: cognitive enhancement, social enhancement, guilt and dependence, and anxiety and arousal. Each item is assessed on a 5-point scale, and scores for each subscale are calculated by averaging across relevant items (i.e., scores on each factor can range from 0-4); higher scores indicate stronger expectancies in that domain.
Incidence of nonmedical prescription stimulant use | 7 months
  Whether or not participants initiate nonmedical prescription stimulant use, and the approximate date, will be assessed over the follow-up period.
Achievement Needs Modification - Self Efficacy for Learning | 7 months
  Achievement needs are being assessed via the Self Efficacy for Learning Form. Items on the Self Efficacy for Learning Form are each scored from 0 - 100 with regard to percent confidence that each behavior can be carried out. Scores across items will be averaged for a total score ranging from 0 to 100, with lower scores indicating poorer self-efficacy and consequently higher achievement needs.
Achievement Needs Modification - Academic Achievement Goals | 7 months
  Achievement needs are also being assessed via the Academic Achievement Goal Questionnaire. A total score will be used for this measure. Each item is answered on a 7 point scale; thus, scores can range from 0 to 72, with higher scores indicating strong achievement goals/needs.

SECONDARY OUTCOMES:
Intention to Use | 7 months
  Intention to engage in nonmedical prescription stimulant use in the following 6 months will be assessed as a proxy of incident of use, and used in analyses if incidence of use is low across all groups. This will be assessed via a 100mm Visual Analogue Scale (0-100). Higher scores indicate higher intention to engage in use.
Modification of Caffeine Expectancy Effects | 7 months
  The Caffeine Expectancy Questionnaire will be used to examine whether expectancy effects for caffeine were modified for the Caffeine-Based Expectancy Challenge group specifically. This measure includes 7 factors, though only Energy/work enhancement, social/mood enhancement, and anxiety/negative physical effects will be analyzed. Items are answered along a 6 point scale (0-5), and scores for each factor are averaged; higher scores indicate stronger expectancies.
Modification of Alcohol Expectancy Effects | 7 months
  The Comprehensive Effects of Alcohol Questionnaire will be used to examine whether expectancy effects for alcohol are modified over time; this is being utilized to ensure that the interventions had specific effects on prescription stimulants and caffeine, and not substance use in general. Positive and negative expectancies can be assessed with this measure, and scores are computed by averaging items loading onto each factor. Items are scored along a 4 point scale (0-3).
Subjective Mood and Arousal | 2 weeks
  Changes in subjective mood and arousal will be assessed across laboratory visits (i.e., to examine whether expectation to receive Adderall and/or ingestion of 200mg caffeine affects subjective mood) using Visual Analogue Scales. Participants will complete scales for the following items: how well do they expect to perform, feeling good, feeling bad, feeling attentive, feeling focused, feeling high, feeling stimulated, feeling motivated, and amount of effort intended to put forth. Each item is measured along a 100mm scale (0-100), with higher scores indicating stronger subjective effects.
Subjective Drug Effects | 2 weeks
  Changes in experienced drug effects will be assessed across laboratory visits (i.e., to examine whether expectation to receive Adderall and/or ingestion of 200mg caffeine affects experienced drug effects) via the Addiction Research Center Inventory. This measure includes 5 subscales: euphoria (scores range from 0-15), dysphoria (scores range from 0-14), intellectual energy and efficiency (scores range from 0-13), amphetamine effects (scores range from 0-11), and sedation (scores range from 0-15). Higher scores indicate stronger experienced drug effects in each domain.
Conners' Continuous Performance Test III | 2 weeks
  The Conners' Continuous Performance Test III will be used to assess changes in attention, impulsivity, and vigilance across laboratory visits. T-scores are provided for each measure. T-scores between 45 and 69 indicate average performance, while scores outside of that range indicate performance difficulties.
Selective Reminding Test | 2 weeks
  The Selective Reminding Test is a measure of learning and memory to assess whether there are differences across laboratory visits. Number of words (out of 12) recalled across 6 trials are tallied for a measure of immediate memory (range: 0-72). Additionally, the number of words recalled across consecutive trials are measured as an index of movement into long term storage (with higher scores indicating better memory; range: 0-72). Long-term memory is also assessed (range: 0-12, with higher scores indicating better memory), as is recognition memory (range: 0-12, with higher scores indicating better memory).
Paced Auditory Serial Addition Test | 2 weeks
  The Paced Auditory Serial Addition Test will be used to assess differences in processing speed and divided attention across laboratory visits. This test includes 4 trials, each of which provides a total correct score out of 25. A total score is computed (0-100), with higher scores indicating better performance.
Stroop Test | 2 weeks
  The Stroop Test will be used to assess differences in selective attention and processing speed across laboratory visits. This test provides reaction time scores for correct trials (smaller scores indicate better performance), as well as percentage of correct trials (out of 100%; higher scores indicate better performance).
Letter-Number Sequencing | 2 weeks
  The Letter-Number Sequencing test will be used to assess differences in working memory across laboratory visits. This test provides a total score correct (range: 0-30), with higher scores indicating better performance.
Verbal Fluency | 2 weeks
  The Verbal Fluency test will be used to assess verbal fluency and information retrieval across laboratory visits. A total score correct is calculated (no maximum score), with higher scores indicating better performance.
Symbol Search | 2 weeks
  The Symbol Search test will be used to assess processing speed across laboratory visits. A total score correct is calculated (range: 0-60), with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Looby, PhD, Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Looby A, Piccorelli AV, Zimmerman L, Falco C, Livingston NR, Akin C, Benton S, Juliano LM. Expectancy for Adderall influences subjective mood and drug effects regardless of concurrent caffeine ingestion: A randomized controlled trial. Psychopharmacology (Berl). 2024 Jan;241(1):109-118. doi: 10.1007/s00213-023-06467-8. Epub 2023 Sep 23. PMID 37740001